CLINICAL TRIAL: NCT05301894
Title: Long-Term, Open-Label Extension Study to Evaluate the Safety and Tolerability of NBI-827104 in Pediatric Subjects With Epileptic Encephalopathy With Continuous Spike-and-Wave During Sleep
Brief Title: Extension Study to Evaluate NBI-827104 in Pediatric Participants With Epileptic Encephalopathy With Continuous Spike-and-Wave During Sleep
Acronym: Steamboat 2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBI-827104-CSWS2025; 2021-006788-11 (EudraCT Number)
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Epileptic Encephalopathy; Continuous Spike and Wave During Sleep
Keywords: Epilepsy; Epileptic Encephalopathy; Neurocrine; NBI-827104; Steamboat 2
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NBI-827104 (Experimental): NBI-827104 administered orally
  Interventions: Drug: NBI-827104

INTERVENTIONS:
Drug: NBI-827104 — T-type calcium channel blocker.

SUMMARY:
The primary objective for this study is to evaluate the long-term safety and tolerability of NBI-827104 in pediatric participants with epileptic encephalopathy with continuous spike-and-wave during sleep (EECSWS).

DETAILED DESCRIPTION:
This study will enroll participants who completed treatment in the Phase 2, multicenter, randomized, double-blind, placebo-controlled, parallel-group Study NBI-827104-CSWS2010 (NCT04625101). Participants who did not participate in Study NBI-827104-CSWS2010 may also be eligible for enrollment.

ELIGIBILITY:
Key Inclusion Criteria:

For participants who enroll directly following the completion of the Study NBI-827104-CSWS2010:

* Completed 12 weeks of treatment in Study NBI-827104-CSWS2010.

For Participants Who Do Not Enroll Directly from or Did Not Participate in Study NBI-827104-CSWS2010:

* Have diagnosis of EECSWS confirmed by the Diagnosis Confirmation Panel (DCP).

Key Exclusion Criteria:

For participants who enroll directly following the completion of the Study NBI-827104-CSWS2010:

* Have developed any other disorder for which the treatment takes priority over treatment of EECSWS or is likely to interfere with study treatment or impair treatment compliance.

For Participants Who Do Not Enroll Directly from or Did Not Participate in Study NBI-827104-CSWS2010:

* Body weight <15 kg at Day 1.
* Clinically relevant findings related to cardiovascular or laboratory parameters at screening as determined by the investigator.
* Presence of relevant neurological disorders other than EECSWS and its underlying conditions as judged by the investigator. Symptomatic conditions underlying EECSWS (for example, neonatal strokes) have to be stable for at least 1 year prior to screening.
* Planned surgical intervention related to structural abnormalities of the brain from screening through the Week 6 Visit.
* Used any active investigational drug other than NBI-827104 in the context of a clinical study within 30 days or 5 half-lives (whichever is longer) before screening or plans to use such an investigational drug (other than NBI-827104) during the study.
* Have developed any other disorder for which the treatment takes priority over treatment of EECSWS or is likely to interfere with study treatment or impair treatment compliance.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
The Occurrence of Serious Treatment-emergent Adverse Events (TEAEs) | Day 1 up to 238 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — Neurocrine Biosciences
Locations (12):
- United States (7):
  - Neurocrine Clinical Site, Orange, California
  - Neurocrine Clinical Site, Aurora, Colorado
  - Neurocrine Clinical Site, Washington D.C., District of Columbia
  - Neurocrine Clinical Site, Miami, Florida
  - Neurocrine Clinical Site, Rochester, Minnesota
  - Neurocrine Clinical Site, Durham, North Carolina
  - Neurocrine Clinical Site, Cleveland, Ohio
- Neurocrine Clinical Site, Dianalund, Denmark
- Spain (2):
  - Neurocrine Clinical Site, Barcelona
  - Neurocrine Clinical Site, Madrid
- Neurocrine Clinical Site, Zurich, Switzerland
- Neurocrine Clinical Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No